CLINICAL TRIAL: NCT01251250
Title: Phase I Clinical Trial of Neem Leaf Extract for the Treatment of Chronic Lymphocytic Leukemia
Brief Title: Azadirachta Indica in Treating Patients With Chronic Lymphocytic Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: lost sponsor support
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 169009; NCI-2010-02103
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Refractory Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Blotting, Western; Gene Expression Profiling; Flow Cytometry; In Situ Hybridization, Fluorescence; neem oil; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral Azadirachta indica once daily on days 1-28. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: laboratory biomarker analysis; Genetic: western blotting; Genetic: gene expression analysis; Other: pharmacological study; Other: flow cytometry; Genetic: fluorescence in situ hybridization; Biological: azadirachta indica; Genetic: reverse transcriptase-polymerase chain reaction

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies
Genetic: western blotting — Correlative studies
  Other Names: Blotting, Western; Western Blot
Genetic: gene expression analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: flow cytometry — Correlative studies
Genetic: fluorescence in situ hybridization — Correlative studies
  Other Names: fluorescence in situ hybridization (FISH)
Biological: azadirachta indica — Given orally
  Other Names: neem; neem tree
Genetic: reverse transcriptase-polymerase chain reaction — Correlative studies
  Other Names: RT-PCR

SUMMARY:
RATIONALE: Azadirachta indica may be an effective treatment for chronic lymphocytic leukemia. PURPOSE: This phase I trial is studying the side effects and best dose of Azadirachta indica in treating patients with chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the lowest dose of neem leaf extract (NLE) with antileukemic effect and acceptable toxicity in patients with chronic lymphocytic leukemia (CLL). II. Establish the safety and toxicity of NLE in patients with CLL. SECONDARY OBJECTIVES: I. Determine the efficacy of NLE in patients with CLL defined as overall clinical response (CR + PR) by the IWCLL criterion. II. To develop a pharmacokinetic/pharmacodynamic model relating neem leaf extract exposure to toxicity and pharmacodynamic endpoints in CLL patients that will allow personalized dosing to target optimal drug exposure. III. To conduct correlative studies. OUTLINE: This is a dose-escalation study. Patients receive oral Azadirachta indica once daily on days 1-28. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a definitive diagnosis of CLL as defined by the IWCLL criteria
* Patients may not have received any prior treatment for management of CLL; (no more than 30 patients with treatment naive disease will be included in this study)
* Patients with advance stage disease (Rai Stage II-IV) may be included in this clinical trial if they refuse to take standard chemotherapeutic regimens
* Patients with relapsed or relapsed/ resistant may be included in this clinical trial if they refuse to take standard chemotherapeutic regimens
* Patients must understand and voluntarily sign an informed consent form
* Have an ECOG Performance Status of =< 2 at study entry
* Able to adhere to the study visit schedule and other protocol requirements
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 10g/dl
* Platelets >= 50,000/mcl
* Total bilirubin within normal institutional limits
* AST (SGOT)/ ALT (SGPT) =< 2.5 X institutional ULN
* Patients of childbearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Trying to conceive, pregnant or breast feeding female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug
* Patients who are consuming other herbals or non-traditional therapies (i.e. green tea extracts and cumin) within the last 4 weeks(28 days) of initiating this clinical study; note: patient must have stopped herbal or other non-traditional therapies for CLL at least 28 days prior to initiating therapy on this study
* Patients with high-risk cytogenetic (del 17p, del 11q) determined by FISH analysis
* Prior organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Lowest clinically active and tolerable dose | After patients have completed at least 2 treatment courses

CONTACTS AND LOCATIONS:
Overall Officials: Asher Chanan-Khan, Principal Investigator — Roswell Park Cancer Institute